CLINICAL TRIAL: NCT04326361
Title: Neonatal Surgeries in India: A Nationwide Survey Among Neonatal and Pediatric Specialists
Brief Title: A Survey of Neonatal Surgery Practices in India
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate professor, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: MMDU/IEC/109P
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Neonatal Disorder
Keywords: Neonatal; Surgery; Neonatal surgery
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Neonatal surgeries — Current practices of neonatal surgeries in India

SUMMARY:
The study will follow a cross-sectional survey design. The target population for the survey was neonatologists, paediatricians, paediatric surgeons and neonatal surgeons treating the newborn infants. The study will be nationwide survey of neonatal specialists regarding the common neonatal surgeries performed in the tertiary care teaching hospital in India. This cross-sectional survey study will commence once the project is approved by DST's Start-up Research Grant (SRG) approval committee and will continue for the period of two years. The protocol of this study was approved by the Institutional Ethics committee of the recognized tertiary care teaching university and will be conducted in accordance with the declaration of Helsinki guideline (Revised) 2013 and Indian Council of Medical Research guidelines 2017.

DETAILED DESCRIPTION:
The survey instrument will be a validated structured survey questionnaire. The content validity of the structured questionnaire will be reported in terms of validity index (CVI), using ratings of item relevance by content experts.1 The content validation of identified items will be executed by the online Delphi method. Initially first round of Delphi survey of contentment validation will be carried out to achieve a consensus of 80% agreement among the identified panel of 10 experts in the field of neonatology will be consulted during the content validation in each round. If not achieved in first round, second round of Delphi survey of contentment validation will be carried out to achieve a consensus of 80% agreement among the identified panel of 10 experts. As more than 10 experts were deemed to be unnecessary, we will not include more than panel of 10 experts in each Delphi survey. The survey instrument will be created on an online survey platform (Survey Monkey). It was evaluated for both face and content validity by the investigators and approved by the experts. The survey will be pilot tested on a group of neonatologists and pediatricians before distribution. The survey will be administered electronically via email along with instructions and a hyperlink to the survey. The participants will be notified of the voluntary nature of participation, confidentiality and non-compensation for participation. Lists of email addresses of neonatologists and neonatal practitioners were assembled by liaising with the Neonatology Chapter of Indian Academy of Pediatrics (IAP Neochap). The invitation will be sent to the 800 neonatologists and pediatricians nationwide in India. To encourage response rates, an additional survey reminder will be emailed 1 week later.Each question will be validated and reported in term of I-CVI. The overall validation of proposed scale with item pool will be reported with S-CVI after the end of each Delphi method of scale validation. S-CVI will be computed by both approaches, universal agreement calculation method (S-CVI/UA) and averaging calculation method (S-CVI/Ave).Lynn recommended that minimum I-CVI of 0.78, in case of 6 to 10 experts and overall the scale should an SCVI/Ave of 0.90 or higher for considered to have excellent content validity.

ELIGIBILITY:
Inclusion Criteria:

* Years of experience, level of neonatal care provided,
* type-severity-number of patients seen monthly (preterm infants, intubation with assisted ventilation, birth asphyxia/hypoxic ischemic encephalopathy), and availability of pediatric subspecialists including neonatal surgeon,
* students pursuing post-graduation in neonatal and Pediatric surgery.

Exclusion Criteria:

* Undergraduate Bachelor of medicine and Bachelor of Surgery (MBBS) students,
* students who are not willing to participate in the study.

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Neonatologists Pediatricians Neonatal and Pediatric surgeons
Sampling Method: Probability Sample
Enrollment: 930 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 1 day (Once through cross-sectional survey)
  Validated structured survey questionnaire will be circulated through SurveyMonkey

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, MPT, Principal Investigator — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Bhatnagar SN, Sarin YK. Current trends in neonatal surgery in India. J Neonatal Surg. 2012 Apr 1;1(2):18. eCollection 2012 Apr-Jun. No abstract available. PMID 26023377
- [Background] Siddharth V, Gupta SK, Agarwala S, Satpathy S, Goel P. Outcome of Care Provided in Neonatal Surgery Intensive Care Unit of a Public Sector Tertiary Care Teaching Hospital of India. J Indian Assoc Pediatr Surg. 2019 Oct-Dec;24(4):257-263. doi: 10.4103/jiaps.JIAPS_177_18. PMID 31571756
- [Background] Lin T, Pimpalwar A. Minimally invasive surgery in neonates and infants. J Indian Assoc Pediatr Surg. 2010 Jan;15(1):2-8. doi: 10.4103/0971-9261.69133. PMID 21180496
- [Result] Puri A, Lal B, Nangia S. A Pilot Study on Neonatal Surgical Mortality: A Multivariable Analysis of Predictors of Mortality in a Resource-Limited Setting. J Indian Assoc Pediatr Surg. 2019 Jan-Mar;24(1):36-44. doi: 10.4103/jiaps.JIAPS_30_18. PMID 30686886
- See also: A Pilot Study on Neonatal Surgical Mortality: A Multivariable Analysis of Predictors of Mortality in a Resource-Limited Setting. — https://www.ncbi.nlm.nih.gov/pubmed/30686886
- See also: Current Trends in Neonatal Surgery in India — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4420385/
- See also: Outcome of Care Provided in Neonatal Surgery Intensive Care Unit of a Public Sector Tertiary Care Teaching Hospital of India. — https://www.ncbi.nlm.nih.gov/pubmed/31571756
- See also: Minimally invasive surgery in neonates and infants — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2998663/